CLINICAL TRIAL: NCT02854865
Title: Feasibility of Speckle Tracking Echocardiography for Estimation of Left Ventricular Filling Pressures in Cardiac Surgery Patients: a Transoesophageal Study
Brief Title: Specke Tracking Echocardiography And Filling Pressures
Acronym: TEE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ulrike Weber, M.D., Medical University of Vienna
Other Study IDs: 1791/2012
Record Dates: First submitted 2016-07-20; First posted 2016-08-04 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Echocardiography, 2-D

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Echocardiography: assess whether GLPSS measured during cardiac surgery using AFI is superior to E/Ea ratio in estimation of LVFP measured as PCWP
  Interventions: Other: echocardiography

INTERVENTIONS:
Other: echocardiography — assess whether GLPSS measured during cardiac surgery using AFI is superior to E/Ea ratio in estimation of LVFP measured as PCWP

SUMMARY:
Determining the LV filling pressure is a key element in the diagnosis and management of patients with suspected decompensated heart failure. The aim of the present study is to assess whether a systolic 2D-STEderived parameter, global longitudinal peak systolic strain (GLPSS), acquired by transoesophageal echocardiography (TEE) is superior to the E/Ea ratio in the estimation of the LVFP measured as the pulmonary capillary wedge pressure (PCWP) in patients during cardiac surgery. Automated function image (AFI) algorithm is a novel method based on 2D strain imaging that enables the simultaneous quantification of myocardial strain in different left ventricular segments; its 3-click method minimizes variability related to a manual training of endocardial border required in an usual 2D-strain analysis.

AFI provides GLPSS by averaging mid-oesophageal 4-, 2- chamber and long axis views. The study is a prospective observational single-center cohort study. 30 Patients scheduled for elective cardiac surgery will be included in the study group. The study is designed to assess whether GLPSS measured during cardiac surgery using AFI is superior to E/Ea ratio in estimation of LVFP measured as PCWP.

DETAILED DESCRIPTION:
For normal cardiac performance, the left ventricle (LV) must be able to eject an adequate stroke volume at arterial pressure (systolic function) and fill without requiring an elevated left atrial (LA) pressure (diastolic function). These systolic and diastolic functions must be adequate to meet the needs of the body. Systolic function is conveniently (although not always accurately) measured as the ejection fraction (EF), calculated as stroke volume divided by end-diastolic volume. Diastolic function has been more difficult to evaluate and is characterized by changed left ventricular (LV) filling dynamics. The mean LA pressure is the source pressure for LV filling. Determining the LV filling pressure is a key element in the diagnosis and management of patients with suspected decompensated heart failure. Measurement of the pulmonary capillary wedge pressure (PCWP) with the Swan-Ganz catheter has become the gold standard for determining LV filling pressure. Invasively measured pulmonary capillary wedge pressure (PCWP) has been widely used as a surrogate for left ventricular filling pressure (LVFP) and is directly associated with functional capacity and prognosis in patients with heart failure. On the other hand, invasive procedures can produce complications, especially in critically ill patients and randomized clinical studies found no benefit from the use of the Swan-Ganz catheter to manage critically ill patients. Thus, efforts to find a noninvasive method of determining LV filling pressure have continued. One of the basic non-invasive parameters which reflect the LVFP is the ratio of peak early diastolic transmitral flow velocity (E) to peak early diastolic velocity of mitral annular motion (Ea) derived from conventional pulsed-wave and Doppler tissue echocardiography. The E/Ea ratio has been found to be superior to individual Doppler tissue imaging (DTI) parameters and to conventional pulsed-wave Doppler parameters assessing LV filling or pulmonary venous flow both in predicting the increase in LVFP and assessing of patient prognosis. However, DTI has inherent limitations which may have a negative impact on the accuracy of Ea measurements. Specifically, DTI is angle-dependent, and is affected by tethering, myocardial translation, and respiration motions. Recently, 2-dimensional speckle tracking echocardiography (2DSTE) has been introduced for the measurement of systolic and diastolic strain and strain rates (SRs) which does not have the above-mentioned limitations. Since most echocardiographic studies evaluating LVFP were performed with transthoracic echocardiography (TTE) in a cardiological setting and primarily diastolic 2D-STE parameters were described, the aim of the present study is to assess whether a systolic 2D-STEderived parameter, global longitudinal peak systolic strain (GLPSS), acquired by transoesophageal echocardiography (TEE) is superior to the E/Ea ratio in the estimation of the LVFP measured as the pulmonary capillary wedge pressure (PCWP) in patients during cardiac surgery. Automated function image (AFI) algorithm is a novel method based on 2D strain imaging that enables the simultaneous quantification of myocardial strain in different left ventricular segments; its 3-click method minimizes variability related to a manual training of endocardial border required in an usual 2D-strain analysis.

AFI provides GLPSS by averaging mid-oesophageal 4-, 2- chamber and long axis views. The study is a prospective observational single-center cohort study. Patients scheduled for elective cardiac surgery will be included in the study group. Written informed consent will be obtained from all patients before surgery. 30 consecutive patients scheduled for elective cardiac surgery who do not meet the exclusion criteria. The study is designed to assess whether GLPSS measured during cardiac surgery using AFI in 45 consecutive patients is superior to E/Ea ratio in estimation of LVFP measured as PCWP.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective cardiac surgery

Exclusion Criteria:

* non-sinus rhythm
* severe mitral regurgitation
* mitral stenosis
* prosthetic mitral valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients schedulded for elective cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
global longitudinal peak systolic strain (GLPSS) acquired by transoesophageal echocardiography | 30min after Induction of anaesthesia
  postoperative offline measurement of strain

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Weber, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical university of vienna, General hospital of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No